CLINICAL TRIAL: NCT01585974
Title: Duration of Treatment With TKIs in the Treatment of Metastatic Renal Cell Carcinoma
Brief Title: Duration of Treatment With Tyrosine Kinase Inhibitors in the Treatment of Metastatic Renal Cell Carcinoma
Acronym: TURCOS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16263; NX1211TR (Other: company internal)
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; TKI; Turkey; Observational
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — All dosage, frequency and duration for drugs will be under the decision of the treating physician

SUMMARY:
This study is a prospective, non-interventional, non-controlled, multi-center, observational cohort study. The medication is prescribed within the regular practice of the physician. Duration and dosage of treatment is solely at the discretion of the attending physician. The primary objective of this study is to assess duration of treatment in Turkish renal cell carcinoma patients treated with TKIs (Tyrosine Kinase Inhibitors) who could not tolerate prior cytokine treatment within the first month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed as metastatic renal cell carcinoma
* Previous cytokine therapy
* To sign informed consent form (ICF)

Exclusion Criteria:

* Patients not willing to sign informed consent form or who withdraw their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as metastatic renal cell carcinoma and could not tolerate previous cytokine therapy within the first month of treatment
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Duration of treatment: from start of tyrosine kinase inhibitor treatment to permanent discontinuation of the product | After 2 years

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAE) | After 2 years
Change of Tumor status | Baseline and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Turkey (Türkiye)

REFERENCES:
- [Derived] Benekli M, Gumus M, Ozkan M, Dane F, Elkiran ET, Cicin I, Sevinc A, Aliustaoglu M, Isikdogan A, Meydan N, Oksuzoglu B, Ozyilkan O, Artac M, Ozdemir F, Kilickap S. Tyrosine kinase inhibitors in the treatment of metastatic renal cell cancer patients with early cytokine intolerance: TURCOS, a Turkish national, prospective observational study. J Oncol Pharm Pract. 2021 Oct;27(7):1623-1630. doi: 10.1177/1078155220963535. Epub 2020 Oct 13. PMID 33050804